CLINICAL TRIAL: NCT02638688
Title: Uterine Fibroid Volume After Myomectomy Compared to Pre-operative Measurement by Two and Three-dimensional Ultrasound
Brief Title: Measurement of Fibroid Volume and 2D, 3D US
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Sherin A Shazly, Faculty, Zagazig University
Other Study IDs: s.shazly; 2011 (Registry Identifier: sherin)
Record Dates: First submitted 2015-12-18; First posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Gynecology
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 2D ultrasound: 2D-US measurements are the most accurate method for measuring fibroid volumes
  Interventions: Other: ultrasound
- 3D ultrasound: 3D-US measurements are the most accurate method for measuring fibroid volumes
  Interventions: Other: ultrasound
- postoperative: actual volume using change in water path measurements are the most accurate method for measuring fibroid volumes
  Interventions: Other: ultrasound

INTERVENTIONS:
Other: ultrasound

SUMMARY:
Objective: To compare 2-dimensional and 3-dimensional ultrasound measurements with the actual myomas volume after surgical removal, to clinically test the validity and usability of 3D ultrasound technology as opposed to conventional 2D real-time ultrasound and to assess the reliability of different ultrasound methods to measure volume of uterine fibroids.

ELIGIBILITY:
Inclusion Criteria:

* surgical intervention

Exclusion Criteria:

* unfit for surgery

Ages: 22 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 44
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2012-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
measuring fibroid volumes | 2012-2015